CLINICAL TRIAL: NCT00247858
Title: Analysis of Methicillin Resistant Staphylococcus Aureus (MRSA) Obtained Through the Emergency Department in a Tertiary Care Hospital in Vancouver Canada From 2001-2005
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Other Study IDs: C05-0247
Record Dates: First submitted 2005-11-01; First posted 2005-11-02 (Estimated); Last update posted 2025-02-11 (Actual); Status verified 2011-09

CONDITIONS: Infection With MRSA Bacteria
Keywords: MRSA, USA300, CMRSA-10, CMRSA-6, soft tissue abscesses

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
To analyze microbiological data from MRSA samples obtained through the emergency department from 2001-2005. There is a strong clinical suspicion that we are now seeing an outbreak of a new strain of MRSA and we plan to better characterize the Vancouver population and complete a chart review to assess specific associated factors.

DETAILED DESCRIPTION:
Pulse field gel electrophoresis, SCC mec typing, antibiotic susceptibilities, presence of the Panton-Valentine Leukocidin gene will be carried out. Clinical manifestations and associated factors will be assessed via chart review. These include: recent antibiotic use, recent hospitalization, IV drug use, HIV status, number of co-morbidities identified, presence of soft tissue abscess, post operative status, presence of bacteremia, residence in Vancouver's downtown eastside (an area of particularly low socioeconomic status).

ELIGIBILITY:
Inclusion Criteria:

* Patient had a microbiological sample submitted from the emergency department of the study hospital from 2001- 2005 which grew MRSA.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a microbiological sample submitted from the emergency department of the study hospital.
Sampling Method: Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2005-01-01; Primary Completion 2012-12-01 (Actual); Study Completion 2012-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Reynolds, MD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada